CLINICAL TRIAL: NCT03883802
Title: A Randomized, Multicentre, Open-Label Controlled Phase II Trial of Foxy-5 as Neo-Adjuvant Therapy in Subjects With Wnt-5a Low Colon Cancer
Brief Title: Foxy-5 as Neo-Adjuvant Therapy in Subjects With Wnt-5a Low Colon Cancer
Acronym: NeoFox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: WntResearch AB (Industry)
Collaborators: SMS-Oncology BV (Unknown); SAGA diagnostics AB (Unknown); Unilabs A/S (Unknown); BioVica AB (Unknown); Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMS-0472B; 2018-003074-27 (EudraCT Number)
Record Dates: First submitted 2018-12-26; First posted 2019-03-21 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Foxy-5 peptide; Folfox protocol

STUDY DESIGN:
Intervention Model Description: two-arm study, 1 to 1 randomization: treatment group and standard therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foxy-5 (Experimental): Arm will receive Foxy-5 as neo-adjuvant therapy prior to surgical removal of tumour and afterwards until initiation of FOLFOX 6 months regimen
  Interventions: Drug: Foxy-5; Drug: FOLFOX regimen; Procedure: Tumour resection (colon cancer surgery)
- Standard therapy (Active Comparator): Surgical removal of tumour followed by 6 months FOLFOX regimen
  Interventions: Drug: FOLFOX regimen; Procedure: Tumour resection (colon cancer surgery)

INTERVENTIONS:
Drug: Foxy-5 — Lyophilized powder for solution for intravenous infusion
  Arms: Foxy-5
Drug: FOLFOX regimen — 6 months treatment regimen
Procedure: Tumour resection (colon cancer surgery) — Surgical removal of patients colon cancer

SUMMARY:
Phase II study investigating the safety, tolerability and effect on disease reccurence of Foxy-5 as neo-adjuvant therapy in resected colon cancer patients treated with FOLFOX chemotherapy regimen. It is a two-arm study and patients will be randomised to receive either standard therapy (surgery + FOLFOX 6 months regimen) or standard therapy + neo-adjuvant administration of Foxy-5 prior to- and following surgery (maximum of 39 administrations) until initiation of FOLFOX therapy.

DETAILED DESCRIPTION:
Foxy-5 is a synthetic hexapeptide with a formylated N-terminus, derived from the protein sequence of the Wnt-5a protein. Low/no expression levels of Wnt-5 protein in primary tumour cells have been correlated to high risk of recurrent metastatic disease and shortened survival in several different types of cancer patients, including colon cancer.

Current standard therapy involves surgical removal of the tumour followed by 6 months treatment with chemotherapy (FOLFOX). Foxy-5 is expected to decrease migration of cancer cells, in subjects with low/absent levels of Wnt-5a protein in their primary tumour and hence result in lower recurrence and a better overall survival. The trial intends to establish the safety and tolerability of Foxy-5 and to evaluate early signs of anti-metastatic activity in subjects with resectable colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to provide written informed consent before any trial-related activities.
2. 18 years of age or older.
3. Male or female subjects with adenocarcinoma of the colon, judged by CT or MRI as either one of the following stages per TNM classification of colon cancer (8th edition, 2017):

   T1-4, N1-2, M0 or T4, N0, M0 and who are considered to fulfil the local criteria for adjuvant post- operative chemotherapy after scheduled surgery.
4. Scheduling of surgery according to local practice allows at least 9 pre- surgery administrations of Foxy-5 for the subject. (Please note: surgery should not be postponed for trial purposes.)
5. Sexually active women of childbearing potential (WOCBP) and males with WOCBP partners who are randomized to the Foxy-5 Arm must use a highly effective method of contraception for the treatment duration and for 28 days after last Foxy-5.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Clinical laboratory values at screening:

   1. Absolute neutrophil count ≥1.5 x 109/L
   2. Haemoglobin ≥ 9 g/dL
   3. Platelets ≥ 100 x 109/L
   4. Aspartate Transaminase (AST) and Alanine Transaminase (ALT)

      ≤1.5x Upper Limit of Normal (ULN)
   5. Serum bilirubin ≤1.5 x the ULN
   6. Creatinine clearance >60 mL/min (determined by Cockcroft-Gault Equation).

Exclusion Criteria:

1. Assessed as not suitable or unable to tolerate adjuvant chemotherapy.
2. Evidence of distant metastatic (M1) disease at Screening (N1-2 is allowed).
3. Any surgery (except tumour biopsy) or therapy with immune suppressive agents or bone marrow stimulating factors within the last two weeks prior to randomization.
4. Any active infection requiring IV antibiotic treatment at the time of screening.
5. History of hematologic or primary solid tumour malignancy.
6. Pregnant or breastfeeding women.
7. Currently participating in another trial and receiving trial therapy or received investigational therapy within 4 weeks of the first dose of Foxy-5.
8. Any other condition or treatment that, in the opinion of the Investigator, might interfere with the trial or current drug or substance abuse.
9. Inability to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial.
10. Unlikely to comply with the protocol requirements, instructions and trial-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial.
11. Legal incapacity or limited legal capacity.
12. Any condition, which results in an undue risk for the subject during the trial participation according to the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of randomization until 28 days after the last dose of Foxy-5, assessed up to 120 days
  The incidence of adverse events (AEs) related to Foxy-5 administration of Grade 3 and higher according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) and the Clavien-Dindo classification of surgical complications. cancer.
ctDNA as surrogate marker for disease free period | 2 years after resection of colon cancer
  The level of ctDNA in plasma of subjects with Wnt-5a low colon cancer as a surrogate parameter for disease recurrence in subjects with Wnt-5a low colon cancer treated with Foxy-5 compared to subjects with Wnt-5a low colon cancer who are in the Control Arm.

SECONDARY OUTCOMES:
Overall survival | 2 years after resection of tumour
  OS at 2 years after resection of the colon cancer
Disease-Free Survival | 2 years after resection of tumour
  DFS at 2 years after resection of the colon cancer
Recurrence-Free Interval | study start to 2 years after resection of tumour
  Recurrence-free interval (RFI) defined as the time from randomization to tumour recurrence.
ctDNA in Wnt-5a high patients | 2 years after resection of tumour
  The level of ctDNA in plasma of subjects with Wnt-5a high colon cancer.

OTHER OUTCOMES:
Thymidine Kinase activity | 1 year after resection of tumour
  The level of thymidine kinase activity in serum in relationship to Wnt- 5a expression in the tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Salazar, MD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Instituto de Investigación Sanitaria INCLIVA, Valencia, Spain